CLINICAL TRIAL: NCT06006442
Title: Vaping-Related Seizures - A Prospective Case-Crossover Study
Brief Title: Vaping-Related Seizures - A Prospective Study
Status: Withdrawn | Type: Observational
Why Stopped: Study was not initiated
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Peter.S.Tatum, Epilepsy Fellow, Dartmouth-Hitchcock Medical Center
Other Study IDs: TatumVRS
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Evaluate the Association of Vaping With Seizures
MeSH Terms: interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DHMC Ambulatory EEG Patients: Dartmouth Hitchcock Medical Center (DHMC) patients aged 21 years or older who already have planned ambulatory EEG study ordered and admit to vaping.
  Interventions: Behavioral: Vaping

INTERVENTIONS:
Behavioral: Vaping — Subjects will be smoking the vapnig products that they admitted to using at baseline in the personal life prior to this study

SUMMARY:
This case-crossover study evaluates the association between vaping and seizures in patients of a large academic medical center who admits to vaping and hav a planned ambulatory EEG ordered.

DETAILED DESCRIPTION:
This case-crossover study will evaluate the short-term effects (seizures) of intermittent exposure to vaping nicotine and/or marijuana products among Dartmouth Hitchcock Medical Center (DHMC) patients aged 21 years or older who already have planned ambulatory EEG study ordered and admit to vaping. The duration of data collection will vary (24-72 hours) depending on ambulatory EEG length was ordered.

Inclusion criteria includes any DHMC patient who admits to vaping and has a planned ambulatory EEG of any duration, regardless of diagnosis or reason for study. Exclusion criteria will include subjectively admitting to using any illicit drugs other than cannabinoids since within 7 days of the study and/or anyone who denies smoking since it would be an ethical issue having someone smoke for the first time during a research study.

All subjects will sign a DHMC and IRB approved consent form to participate in the study before it starts. They will receive one copy and another copy will be kept by DHMC in the patient chart. An optional survey/questionnaire will be obtained before the study to confirm if the patient vapes, what products and doses they use, and what other medications or drugs they use. Personal information will also be obtained for later stratification, including age, sex, sexuality, household income, race, ethnicity, heritage, culture, education level, medical history, psychiatric history.

During the study, subjects will keep a vaping diary for 24 to 72 hours depending on how long their study was ordered for. All patients will document the dates, times, contents, brands, sources, doses, and durations of use in their vaping diary which will be handed to the research team at the end of the study.

Each patient will serve as their own control by assessing EEG for seizures and interictal discharges at different times as follows:

* A 60-minute period starting 60 minutes prior to the start of a vaping event which was associated with a seizure.
* A 30-minute period starting 8 hours prior to the start of a vaping event which was associated with a seizure.
* A 30-minute period starting 24 hours prior to the start of a vaping event which was associated with a seizure.
* A 30-minute period randomly selected during a time that no seizures objectively occurred on EEG

During the analysis phase of the study, data will be stratified for age, sex, race, ethnicity, current socio-economic status, prescription medications with known epileptogenic side effects, prior diagnosis of psychogenic non-epileptic seizures, prior psychiatric diagnoses, and prior poly-substance with a negative drug test at time of study.

Outcome measures will include the odds of having seizures or interictal discharges during the 4 control times will be calculated and compared to the odds of experiencing a seizure or interictal discharge within the hypothesized one hour after completing vaping. The quantitative outcome will be odds ratios.

There is no risk put placed on patients in this study since they are using vaping products without alteration from their daily life.

EEG data will be obtained from DHMC epilepsy patients through the NATUS system. Data will be stored in the patient's electronic medical record system at DHMC. Only members of the epilepsy team at DHMC will have access to this password protected research data which will include: EEG recordings, patient and staff member journal entry, pre-study survey, EDH note, Signed consent

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria includes any DHMC patient who admits to vaping and has a planned ambulatory EEG of any duration, regardless of diagnosis or reason for study.

Exclusion Criteria:

* Exclusion criteria will include subjectively admitting to using any illicit drugs other than cannabinoids since within 7 days of the study and/or anyone who denies smoking since it would be an ethical issue having someone smoke for the first time during a research study.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any DHMC patient aged 21 years or above with a planned ambulatory electroencephalogram (EEG) of any duration, regardless of diagnosis or reason for study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Odds of Vaping Related Seizure | The hour before and after vaping, 8 hours prior to vaping, and 24 hours prior to vaping
  Odds ratio of vaping during periods of seizures versus periods of seizure freedom.

SECONDARY OUTCOMES:
Odds of Increased Interictal Discharges After Vaping | The hour before and after vaping, 8 hours prior to vaping, and 24 hours prior to vaping
  Odds ratio of vaping during periods of increased epileptiform discharges compared to normal baseline EEG background.

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Tatum, DO, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided